CLINICAL TRIAL: NCT03058510
Title: Feasibility of Orbital Atherectomy System in Calcified Bifurcation Lesion
Acronym: ORBID-OA
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: GCO 16-1561
Record Dates: First submitted 2017-02-16; First posted 2017-02-23 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Coronary Artery Disease
Keywords: bifurcation lesion; atherectomy; calcification; stent
MeSH Terms: conditions — Coronary Artery Disease; Calcinosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stable CAD Patients: Stable CAD patients with calcified bifurcation lesion
  Interventions: Procedure: Frequency domain optical coherence tomography

INTERVENTIONS:
Procedure: Frequency domain optical coherence tomography — OCT is an established medical imaging technique that uses light to capture high-resolution, three-dimensional images of blood vessels
  Other Names: coronary angiogram; FD OCT

SUMMARY:
ORBID-OA is a single-center, observational study in 30 patients with stable coronary artery disease.

The aim of the study is to analyze the outcomes of main vessel stenting on side branch in calcified bifurcation lesion and identify preprocedural predictors of side branch complication by utilizing two-dimensional (2D) and three-dimensional (3D) frequency domain optical coherence tomography (FD-OCT).

DETAILED DESCRIPTION:
Coronary artery bifurcation lesion is a common lesion subset in PCI accounting for 15-20% of the total number of interventions (1). Treatment of coronary artery bifurcation lesions represents a challenging area in interventional cardiology (2). When compared with non-bifurcation interventions, bifurcation interventions have a lower rate of procedural success, higher procedural costs, longer hospitalization and a higher clinical and angiographic restenosis (3). Factors contributing to this adverse outcome include limitations of angiography in assessment of side-branch (SB) disease severity and the lack of established angiographic predictors of SB patency and lumen compromise. Better understanding of the underlying plaque morphology and plaque composition may facilitate more effective treatment of bifurcation lesions.

Heavy calcification within coronary atherosclerotic plaque adversely influences both clinical and procedural success after percutaneous coronary interventions (PCI) (4,5). The use of drug-eluting stent (DES) in calcified lesions poses special challenges. Atherectomy can facilitate successful stent delivery and expansion in calcified lesions. Orbital atherectomy (OA) is the newly FDA approved device for treatment of severely calcified coronary lesions which works on the principle of elliptical burr movement. The ORBIT I and II clinical trials evaluated the safety of OA in de novo calcified coronary lesions and demonstrated that complication rate was comparable to historical controls of rotational atherectomy (6).

Intravascular imaging has provided new understanding of mechanisms associated with SB compromise following bifurcation PCI (7-9). Plaque shift has been traditionally considered as the principal mechanism for side-branch compromise after main vessel intervention (9), however recent intravascular imaging studies have provided new insights by suggesting carina shift as a major mechanism implicated in side-branch closure (7). Intravascular ultrasound (IVUS) has been used for guidance in bifurcation lesions, aiding the visualization of plaque morphology at the main vessel and the side-branches and helping the selection of stent size and length as well as the selection of stenting strategy. However, due to the low spatial resolution of IVUS, all attempts for three-dimensional visualization have only focused on visualization of the luminal contour and not on the vessel morphology or the vessel-stent interaction. Optical coherence tomography (OCT) has ~10 times higher resolution than IVUS which allows precise evaluation of the microstructure of the vessel wall including lipid pool, fibrous cap, calcification, and thrombus (10). In addition, it provides immediate automated measurements for lumen dimensions before the treatment and precise evaluation of strut apposition and stent expansion after stenting, which is of particular interest in bifurcation PCI, since it's been associated with a higher number of malapposed stent struts and more frequent stent underexpansion leading to higher incidence of stent thrombosis and restenosis.

OCT has been shown to constitute a valuable tool for PCI guidance and also the utility of three-dimensional (3D) renderings for assessing the mechanism of side-branch compromise following intervention in bifurcation lesions. (11,12). The recent development of OCT with online 3D reconstruction allows the operator to obtain a 3D visualization of the lesion and may provide a unique tool for guidance during complex bifurcation PCI and potentially improve stenting results (12). 3D OCT has been used to visualize jailed side branches after implantation of bioresorbable scaffolds in the main branch and develop a new classification system based on the number of SB compartments (13). In addition, its potential clinical application in guiding the rewiring of the distal compartment of the SB ostium (jailed with stent struts after MB stenting) to minimize the risk of floating struts was demonstrated.

The aim of the study is to analyze the outcomes of main vessel stenting on side branch in calcified bifurcation lesion and identify preprocedural predictors of side branch complication by utilizing two-dimensional (2D) and three-dimensional (3D) frequency domain optical coherence tomography (FD-OCT). Thirty consecutive patients with calcified lesions requiring PCI of main vessel with drug eluting stent implantation for the treatment of stable CAD will be included in the study. All potential subjects will sign a separate Mount Sinai surgical/procedure informed consent for their Cardiac Catheterization procedure on the day of their hospital visit.

Patients will undergo coronary angiogram. OCT will be performed to analyze plaque morphology, the extent and location of calcification, side branch size, angle, and ostial involvement. Patients will undergo PCI with stent implantation according to current standards of care. Lesion preparation including lesion pre-dilation, and use of atherectomy and protection devices will be performed at the operator's discretion, followed by MV stenting. The operator will also decide on length and size of the implanted stent. Procedural optimization, such as post-dilation or additional stent implantation will be performed based only on the angiographic findings, according to the discretion of the operator. Coronary angiogram and another OCT pullback will be performed after PCI.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 years of age presenting with stable coronary artery disease.
* Angiographic lesion with severe calcification with or without side branch (SB) in whom provisional main vessel stenting strategy is planned after reviewing angiogram will be recruited

Exclusion Criteria:

* Patients with ostial left main artery lesions or ostial right coronary artery lesions
* Female patients with child bearing potential not taking adequate contraceptives or currently breastfeeding
* Known allergy to acetylsalicylic acid or clopidogrel.
* Planned surgery within 12 months.
* History of bleeding diathesis
* Major surgery within 15 days
* Life expectancy < 12 months.
* Patients with kidney dysfunction (CrCl<30)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thirty consecutive patients with calcified lesions requiring PCI of main vessel with drug eluting stent implantation for the treatment of stable CAD will be included in the study.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-01-17 (Actual); Primary Completion 2017-10-13 (Actual); Study Completion 2017-10-13 (Actual)

PRIMARY OUTCOMES:
Procedural success | Day 1
  Incidence of placing a stent with less than 50% residual stenosis

SECONDARY OUTCOMES:
Acute angiographic complications | Day 1
  Incidence of acute angiographic complications

CONTACTS AND LOCATIONS:
Overall Officials: Annapoorna Kini, MD MRCP FACC, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai and the Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al Suwaidi J, Berger PB, Rihal CS, Garratt KN, Bell MR, Ting HH, Bresnahan JF, Grill DE, Holmes DR Jr. Immediate and long-term outcome of intracoronary stent implantation for true bifurcation lesions. J Am Coll Cardiol. 2000 Mar 15;35(4):929-36. doi: 10.1016/s0735-1097(99)00648-8. PMID 10732890
- [Background] Iakovou I, Ge L, Colombo A. Contemporary stent treatment of coronary bifurcations. J Am Coll Cardiol. 2005 Oct 18;46(8):1446-55. doi: 10.1016/j.jacc.2005.05.080. Epub 2005 Sep 28. PMID 16226167
- [Background] Sharma SK, Sweeny J, Kini AS. Coronary bifurcation lesions: a current update. Cardiol Clin. 2010 Feb;28(1):55-70. doi: 10.1016/j.ccl.2009.10.001. PMID 19962049
- [Background] Writing Group Members; Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, Das SR, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Isasi CR, Jimenez MC, Judd SE, Kissela BM, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Magid DJ, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Rosamond W, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee; Stroke Statistics Subcommittee. Executive Summary: Heart Disease and Stroke Statistics--2016 Update: A Report From the American Heart Association. Circulation. 2016 Jan 26;133(4):447-54. doi: 10.1161/CIR.0000000000000366. No abstract available. PMID 26811276
- [Background] Moussa I, Ellis SG, Jones M, Kereiakes DJ, McMartin D, Rutherford B, Mehran R, Collins M, Leon MB, Popma JJ, Russell ME, Stone GW. Impact of coronary culprit lesion calcium in patients undergoing paclitaxel-eluting stent implantation (a TAXUS-IV sub study). Am J Cardiol. 2005 Nov 1;96(9):1242-7. doi: 10.1016/j.amjcard.2005.06.064. Epub 2005 Sep 15. PMID 16253590
- [Background] Parikh K, Chandra P, Choksi N, Khanna P, Chambers J. Safety and feasibility of orbital atherectomy for the treatment of calcified coronary lesions: the ORBIT I trial. Catheter Cardiovasc Interv. 2013 Jun 1;81(7):1134-9. doi: 10.1002/ccd.24700. Epub 2013 Mar 5. PMID 23460596
- [Background] Karanasos A, Tu S, van der Heide E, Reiber JH, Regar E. Carina shift as a mechanism for side-branch compromise following main vessel intervention: insights from three-dimensional optical coherence tomography. Cardiovasc Diagn Ther. 2012 Jun;2(2):173-7. doi: 10.3978/j.issn.2223-3652.2012.04.01. No abstract available. PMID 24282711
- [Background] Suarez de Lezo J, Medina A, Martin P, Novoa J, Suarez de Lezo J, Pan M, Caballero E, Melian F, Mazuelos F, Quevedo V. Predictors of ostial side branch damage during provisional stenting of coronary bifurcation lesions not involving the side branch origin: an ultrasonographic study. EuroIntervention. 2012 Feb;7(10):1147-54. doi: 10.4244/EIJV7I10A185. PMID 22030298
- [Background] Farooq V, Serruys PW, Heo JH, Gogas BD, Okamura T, Gomez-Lara J, Brugaletta S, Garcia-Garcia HM, van Geuns RJ. New insights into the coronary artery bifurcation hypothesis-generating concepts utilizing 3-dimensional optical frequency domain imaging. JACC Cardiovasc Interv. 2011 Aug;4(8):921-31. doi: 10.1016/j.jcin.2011.06.004. PMID 21851908
- [Background] Tearney GJ, Regar E, Akasaka T, Adriaenssens T, Barlis P, Bezerra HG, Bouma B, Bruining N, Cho JM, Chowdhary S, Costa MA, de Silva R, Dijkstra J, Di Mario C, Dudek D, Falk E, Feldman MD, Fitzgerald P, Garcia-Garcia HM, Gonzalo N, Granada JF, Guagliumi G, Holm NR, Honda Y, Ikeno F, Kawasaki M, Kochman J, Koltowski L, Kubo T, Kume T, Kyono H, Lam CC, Lamouche G, Lee DP, Leon MB, Maehara A, Manfrini O, Mintz GS, Mizuno K, Morel MA, Nadkarni S, Okura H, Otake H, Pietrasik A, Prati F, Raber L, Radu MD, Rieber J, Riga M, Rollins A, Rosenberg M, Sirbu V, Serruys PW, Shimada K, Shinke T, Shite J, Siegel E, Sonoda S, Suter M, Takarada S, Tanaka A, Terashima M, Thim T, Uemura S, Ughi GJ, van Beusekom HM, van der Steen AF, van Es GA, van Soest G, Virmani R, Waxman S, Weissman NJ, Weisz G; International Working Group for Intravascular Optical Coherence Tomography (IWG-IVOCT). Consensus standards for acquisition, measurement, and reporting of intravascular optical coherence tomography studies: a report from the International Working Group for Intravascular Optical Coherence Tomography Standardization and Validation. J Am Coll Cardiol. 2012 Mar 20;59(12):1058-72. doi: 10.1016/j.jacc.2011.09.079. Erratum In: J Am Coll Cardiol. 2012 May 1;59(18):1662. Dudeck, Darius [corrected to Dudek, Darius]; Falk, Erlin [corrected to Falk, Erling]; Garcia, Hector [corrected to Garcia-Garcia, Hector M]; Sonada, Shinjo [corrected to Sonoda, Shinjo]; Troels, Thim [corrected to Thim, Troels]; van Es, Gerrit-Ann [correct. PMID 22421299
- [Background] Di Mario C, Iakovou I, van der Giessen WJ, Foin N, Adrianssens T, Tyczynski P, Ghilencea L, Viceconte N, Lindsay AC. Optical coherence tomography for guidance in bifurcation lesion treatment. EuroIntervention. 2010 Dec;6 Suppl J:J99-J106. doi: 10.4244/EIJV6SUPJA16. PMID 21930500
- [Background] Karanasos A, Tu S, van der Linden M, van Weenen S, Ligthart J, Regar E. Online 3-dimensional rendering of optical coherence tomography images for the assessment of bifurcation intervention. Can J Cardiol. 2012 Nov-Dec;28(6):759.e1-3. doi: 10.1016/j.cjca.2012.04.017. Epub 2012 Jul 3. PMID 22763361